CLINICAL TRIAL: NCT02296268
Title: Stepping up Aerobic Exercise to Improve Health Outcomes After Stroke: Translating Research Into Clinical Care
Brief Title: Stepping up Aerobic Exercise to Improve Health Outcomes After Stroke
Acronym: STROKE-TRIC
Status: Completed | Type: Observational
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Principal Investigator, Marilyn MacKay-Lyons, Affiliated Scientist, Nova Scotia Health Authority
Other Study IDs: CDHA-RS 2015-223
Record Dates: First submitted 2014-11-14; First posted 2014-11-20 (Estimated); Last update posted 2018-03-23 (Actual); Status verified 2018-03

CONDITIONS: Stroke
Keywords: stroke; aerobic exercise; screening; prescription
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Pre-Clinic Stroke Group: In- or out-patients with diagnosis of ischemic or hemorrhagic stroke who have been referred to the NSRC prior to the establishment of the Clinic and are willing/able to provide written informed consent and have no contraindications to exercise testing. Utilization of aerobic exercise will be monitored during their physiotherapy sessions (Aim 3).
  Interventions: Behavioral: Aerobic Exercise Screening and Prescription Clinic
- Post-Clinic Stroke Group: In- or out-patients with diagnosis of ischemic or hemorrhagic stroke who have been referred to the NSRC after the establishment of the Clinic and are willing/able to provide written informed consent and have no contraindications to exercise testing. Each patient will undergo an assessment in the Aerobics Clinic and will receive a prescription for aerobic training based on the assessment findings. Utilization of aerobic exercise will be monitored during their physiotherapy sessions (Aim 3).
  Interventions: Behavioral: Aerobic Exercise Screening and Prescription Clinic
- Stroke Rehabilitation Physiotherapists: Physiotherapists whose current practice involves working full-time or part-time on in- or out-patient stroke service at the NSRC. Their self-efficacy regarding the clinical utilization of aerobic exercise post-stroke will be conducted prior to, and after, implementation of the Aerobics Clinic.

INTERVENTIONS:
Behavioral: Aerobic Exercise Screening and Prescription Clinic — Patients will be referred to the Clinic by their physiotherapist to be assessed regarding their safety and readiness to participate in aerobic training. If they are deemed to be safe and ready, an aerobic exercise prescription will be written to guide the implementation of a safe and effective training protocol. Patients deemed to be at moderate to high risk will need to be cleared for testing by a physician on the stroke service. A cardiologist will be consulted about specific concerns re cardiac status.
  Groups: Post-Clinic Stroke Group; Pre-Clinic Stroke Group

SUMMARY:
Stroke is a leading cause of chronic disability here in Nova Scotia and globally. Aerobic exercise is known to improve health by increasing energy levels, physical mobility, balance, bone health, cardiovascular risk reduction, mental well-being, cognition, sleep, and quality of life. Nonetheless, people remain woefully inactive after stroke, regardless if they are in hospital or at home. The current investigative team and others have shown that even during physiotherapy, exercise intensity is not adequate to increase physical fitness. Consequently, patients are often deprived of a treatment that could improve their recovery. Why does this gap between evidence and clinical practice persist? Through a national survey the current team found that an important contributing factor is lack of appropriate screening (especially stress tests) to ensure that patients are safe to engage in aerobic exercise. This project is designed to close this evidence-practice gap by establishing a state-of-the-art aerobic exercise screening and prescription clinic at the Nova Scotia Rehabilitation Centre (NSRC). The intent is to compare outcomes of stroke rehabilitation participants before and after the clinic is underway and determine if the clinic has a positive effect on the confidence of NSRC physiotherapists to use aerobic exercise safely and effectively in stroke rehabilitation.

DETAILED DESCRIPTION:
Research question: To what extent does an on-site aerobic exercise screening and prescription clinic effect uptake of aerobic exercise and patient outcomes in in-patient stroke rehabilitation?

Design: Pre-post cohort design to explore real-world application and feasibility

Aim 1. Establish an aerobic exercise screening and prescription clinic (herein 'Aerobics Clinic') at the NSRC.

Aim 2. Assess the potential impact of the Aerobics Clinic on the self-efficacy of physiotherapists at NSRC regarding clinical utilization of aerobic exercise in in-patient stroke rehabilitation.

Method: An assessment of the physiotherapy participants' self-efficacy regarding the clinical utilization of aerobic exercise post-stroke will be conducted prior to, and after, implementation of the Clinic.

Aim 3: Assess the potential impact of the Aerobics Clinic on prescription and treatment practices regarding aerobic exercise among patients in stroke rehabilitation at the NSRC.

Method: Prior to, and after, implementation of the Clinic the actual utilization of aerobic exercise in the practices of the physiotherapy participants will be assessed using heart rate monitoring, activity monitoring, and health record review.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults
* Diagnosed with ischemic or hemorrhagic stroke
* Referred to NSRC for stroke rehabilitation

Exclusion Criteria:

* Have contraindications to exercise testing using American College of Sports Medicine guidelines

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients post-stroke
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2016-01-30 (Actual); Primary Completion 2018-01-26 (Actual); Study Completion 2018-01-26 (Actual)

PRIMARY OUTCOMES:
Change from admission 6-Minute Walk Test at discharge | admission and discharge (baseline and 5-6 weeks later)
  To assess change between admission and discharge in distance walked without manual support in 6 minutes

SECONDARY OUTCOMES:
Change from admission 10-Meter Walk at discharge | admission and discharge (baseline and ~5-6 weeks later)
  To assess change between admission and discharge in n walking speed over a 10-metre distance
Change from admission resting blood pressure at discharge | admission and discharge (baseline and 5-6 weeks later)
  To assess change between admission and discharge in resting systolic and diastolic blood pressure
Change from admission abdominal girth at discharge | admission and discharge
  To assess change between admission and discharge in waist circumference in relaxed standing position
Change from admission Stroke-Specific Quality of Life at discharge | admission and discharge (baseline and 5-6 weeks later)
  To assess change between admission and discharge in quality of life questionnaire
Change from admission Readiness for Physical Activity Scale at discharge | admission and discharge (baseline and 5-6 weeks later)
  To assess change between admission and discharge in readiness to engage in physical activity
Change from admission Fatigue Severity Scale at discharge | admission and discharge (baseline and 5-6 weeks later)
  To assess change between admission and discharge in level of fatigue

CONTACTS AND LOCATIONS:
Locations (1):
- QEII Health Sciences Centre, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No
We plan to disseminate the findings through a peer-reviewed publication.